CLINICAL TRIAL: NCT01068808
Title: The Development of Allergic Rhinitis in Children Previously Diagnosed as Nonallergic Rhinitis
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Orathai Piboonpocanun, Department of Pediatrics, Faculty of medicine, Siriraj hospital, Mahidol University
Other Study IDs: 640/2552(EC4)
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Allergic Rhinitis (Disorder)
Keywords: Nonallergic rhinitis; Allergic rhinitis; Development
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Patch Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Nonallergic rhinitis: Nonallergic rhinitis (negative skin prick test)
  Interventions: Procedure: skin prick test

INTERVENTIONS:
Procedure: skin prick test — skin prick test to aeroallergen
  Other Names: SPT

SUMMARY:
The purpose of this study is to evaluate development of allergic rhinitis in children with nonallergic rhinitis.

DETAILED DESCRIPTION:
Rhinitis is a common condition associated with significant effects on quality of life. Rhinitis may be divided into two groups, those with concurrent allergy (allergic rhinitis, AR) and those without allergy but who still suffer from nasal symptoms (nonallergic rhinitis, NAR).

Evidence indicated that adult with NAR can have de novo sensitization to aeroallergen (24%), suggesting that patients with NAR might evolve to AR. Thus the purpose of this study is to evaluate development of allergic rhinitis in children with nonallergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Children between the age of 1 year and 15 years with the diagnosis of nonallergic rhinitis who are attending the pediatric allergy clinic during Jan 2005 - Dec 2007.

Exclusion Criteria:

* Patients who have allergic rhinitis and underlying disease eg.chronic renal disease, liver disease, heart disease, cancer.

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The patient from pediatric allergy clinic will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the development of AR in children who were previously diagnosed with NAR | 24 months

SECONDARY OUTCOMES:
To determine the persistence and severity of the symptoms, new comorbidities and triggering factors in children with nonallergic rhinitis | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Orathai Piboonpocanun, Assoc.Prof., Principal Investigator — Division of Allergy and Immunology, Department of Pediatrics, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand
Locations (1):
- Division of Allergy and Immunology, Department of Pediatrics, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Result] Veskitkul J, Vichyanond P, Visitsunthorn N, Jirapongsananuruk O. The development of allergic rhinitis in children previously diagnosed as nonallergic rhinitis. Am J Rhinol Allergy. 2013 Jan;27(1):43-7. doi: 10.2500/ajra.2013.27.3839. PMID 23406600